CLINICAL TRIAL: NCT02930655
Title: A Single-center, Open-label, Randomized, Versus a Control Group, Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Oral Lucerastat in Adult Subjects With Fabry Disease Receiving Enzyme Replacement Therapy
Brief Title: A Study to Assess the Safety and Tolerability of Lucerastat in Subjects With Fabry Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-069-104
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Fabry Disease
Keywords: Fabry disease; lucerastat
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; Enzyme Replacement Therapy; agalsidase beta; agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lucerastat group (Experimental): Ten subjects with Fabry Disease received 1000 mg of oral lucerastat twice daily for 12 weeks in addition to their standard of care treatment (enzyme replace therapy).
  Interventions: Drug: Lucerastat; Drug: Enzyme replacement therapy (ERT)
- Control group (Experimental): Four subjects with Fabry Disease under enzyme replace therapy (ERT) as standard of care treatment were included as a control group.
  Interventions: Drug: Enzyme replacement therapy (ERT)

INTERVENTIONS:
Drug: Lucerastat — Hard gelatin capsules for oral administration formulated at a strength of 250 mg, and administered as 4 capsules in the morning and 4 capsules in the evening.
  Other Names: ACT-434964
  Arms: Lucerastat group
Drug: Enzyme replacement therapy (ERT) — All the subjects received an ERT as background therapy for at least 24 months prior to the screening visit and they had to continue receiving this treatment during the conduct of the study.
  Other Names: Fabrazyme; Replagal

SUMMARY:
The primary purpose of this study was to assess the safety and tolerability of lucerastat in adults with Fabry Disease receiving Enzyme Replacement Therapy (ERT).

The secondary objectives were to investigate the effects of lucerastat on plasma and urine levels of biomarkers, to assess its effects on renal and cardiac functions and to determine the pharmacokinetic profile of lucerastat at steady-state.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Male and female adult subjects with a diagnosis of Fabry Disease (FD) based on historical assessments (residual α-GAL A activity level below lower limit of normal for males and presence of a galactosidase alpha mutation for females) and a history of clinical symptoms of FD
* On ERT for at least 24 months without any change in dose within the last 6 months prior to screening

Exclusion Criteria:

* Severe renal function impairment
* Severe residual neurologic deficit
* Clinically significant unstable cardiac disease
* Any circumstances or conditions, which, in the opinion of the investigator, may have affected full participation in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood pressure | Up to Week 12
Change from baseline in heart rate | Up to Week 12
Change from baseline in electrocardiogram (ECG) variables | Up to Week 12
  The duration (in ms) of the different ECG variables were measured using a standard 12-lead ECG
Change from baseline in body weight | Up to Week 12
Number of subjects with treatment-emergent adverse events and serious adverse events | Up to Week 12
Number of subjects with adverse events leading to premature discontinuation of lucerastat or ERT | Up to Week 12
Number of subjects with treatment-emergent abnormalities in laboratory variables | Up to Week 12

SECONDARY OUTCOMES:
Change from baseline in plasma biomarkers of Fabry Disease | Up to Week 12
  Biomarkers reflecting glycolipid metabolism were measured (unit of measure: ng/mL)
Change from baseline in urine biomarker of Fabry Disease | Up to Week 12
  Biomarker reflecting glycolipid metabolism was measured (unit of measure: ng/mg)
Change from baseline in left ventricular ejection fraction (LVEF) | Up to Week 12
  LVEF was used to monitor cardiac function in subjects with Fabry Disease
Change from baseline in left ventricular mass index (LVMi) | Up to Week 12
  LVMi was used to monitor cardiac function in subjects with Fabry Disease
Change from baseline in estimated glomerular filtration rate (eGFR) | Up to Week 12
  eGFR was used to monitor renal function in subjects with Fabry Disease
Change from baseline in urine albumin-to-creatinine ratio (UACR) | Up to Week 12
  UACR was used to monitor renal function in subjects with Fabry Disease
Maximum plasma concentration (Cmax) of lucerastat | At Week 4 visit, blood samples drawn at the following time points: pre-dose, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 10h, 12h post-dose
  Cmax was determined directly from the observed plasma concentration-time curves of lucerastat. Blood samples for PK analyses were drawn at scheduled time points at the Week 4 visit
Time to reach Cmax (tmax) of lucerastat | At Week 4 visit, blood samples drawn at the following time points: pre-dose, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 10h, 12h post-dose
  tmax was determined directly from the observed plasma concentration-time curves of lucerastat. Blood samples for PK analyses were drawn at scheduled time points at the Week 4 visit
Area under the plasma concentration-time curve [AUC(tau)] of lucerastat | At Week 4 visit, blood samples drawn at the following time points: pre-dose, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 10h, 12h post-dose
  AUC(tau) corresponds to the area under the plasma concentration time curve of lucerastat over a dosing interval (tau = 12 hours)
Terminal half-life [t(1/2)]of lucerastat | At Week 4 visit, blood samples drawn at the following time points: pre-dose, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 10h, 12h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guérard, Study Director — Actelion
Locations (1):
- Investigator Site, Würzburg, Germany

REFERENCES:
- [Derived] Guerard N, Morand O, Dingemanse J. Lucerastat, an iminosugar with potential as substrate reduction therapy for glycolipid storage disorders: safety, tolerability, and pharmacokinetics in healthy subjects. Orphanet J Rare Dis. 2017 Jan 14;12(1):9. doi: 10.1186/s13023-017-0565-9. PMID 28088251